CLINICAL TRIAL: NCT00217503
Title: Primary Effusion Lymphoma: A Pilot Trial of Bevacizumab and Modified Dose-Adjusted Infusional CDE Chemotherapy Preceded by a Brief Pre-Phase Assessment of Targeted Oncolytic Virotherapy With Bortezomib, Zidovudine and Valganciclovir
Brief Title: Bortezomib and Antiviral Therapy Followed By Effusion Drainage, Bevacizumab, and Combination Chemotherapy in Treating Patients With Primary Effusion Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000441214; NCI-05-C-0203; NCI-P6330; NCT00121576 (obsolete NCT alias)
Record Dates: First submitted 2005-09-20; First posted 2005-09-22 (Estimated); Last update posted 2013-06-20 (Estimated); Status verified 2007-04

CONDITIONS: Lymphoma
Keywords: AIDS-related peripheral/systemic lymphoma
MeSH Terms: conditions — Lymphoma | interventions — Bevacizumab; Filgrastim; pegfilgrastim; Bortezomib; Cyclophosphamide; Doxorubicin; Etoposide; Ganciclovir; Valganciclovir; Zidovudine

INTERVENTIONS:
Biological: bevacizumab
Biological: filgrastim
Biological: pegfilgrastim
Drug: bortezomib
Drug: cyclophosphamide
Drug: doxorubicin hydrochloride
Drug: etoposide
Drug: ganciclovir
Drug: valganciclovir
Drug: zidovudine

SUMMARY:
RATIONALE: Herpesvirus is found in the cancer cells of patients with primary effusion lymphoma. Antiviral drugs, such as zidovudine and valganciclovir, may be able to act against the herpesvirus in the cancer cells to help kill the cancer cells. Bortezomib may help the antiviral drugs kill the cancer cells. Draining the effusion removes fluid that has built up. Monoclonal antibodies, such as bevacizumab, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or carry cancer-killing substances to them. Bevacizumab may also stop the growth of cancer cells by blocking blood flow to the cancer. Drugs used in chemotherapy, such as cyclophosphamide, doxorubicin, and etoposide, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving bortezomib together with antiviral therapy followed by effusion drainage, bevacizumab, and combination chemotherapy may kill more cancer cells.

PURPOSE: This phase II trial is studying how well giving bortezomib together with antiviral therapy followed by effusion drainage, bevacizumab, and combination chemotherapy works in treating patients with primary effusion lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the complete response rate in patients with previously untreated primary effusion lymphoma treated with effusion drainage and bevacizumab in combination with chemotherapy comprising cyclophosphamide, doxorubicin, and etoposide.

Secondary

* Determine the overall survival, disease-free survival, and progression-free survival of patients treated with this regimen.
* Determine the toxicity of this regimen in previously treated or untreated patients.
* Determine, preliminarily, the biologic effects of targeted oncolytic virotherapy comprising bortezomib, zidovudine, and valganciclovir in these patients.

OUTLINE: This is a 2-part, pilot study.

Patients who are HIV-positive receive highly-active antiretroviral therapy during study treatment.

* Part 1 (targeted oncolytic virotherapy)*: Patients receive bortezomib IV over 3-5 seconds on days 1, 4, and 8, zidovudine IV over 1 hour twice daily on days 1-10, and oral valganciclovir (or ganciclovir IV) twice daily on days 1-14. One day after completion of zidovudine, patients begin treatment in part 2.

NOTE: *Part 1 treatment may be omitted in patients who are acutely ill with primary effusion lymphoma at study entry AND a 10- to 14-day delay of starting part 2 treatment may pose a hazard to the patient.

* Part 2

  * Effusion drainage: Patients undergo effusion drainage prior to each course of bevacizumab* and chemotherapy. The drainage tube may remain in place to allow for continuous drainage of effusion during treatment with bevacizumab* and chemotherapy.
  * Bevacizumab* plus cyclophosphamide, doxorubicin, and etoposide (iCDE): Patients receive bevacizumab* IV over 30-90 minutes on days 1 and 6, cyclophosphamide, doxorubicin, and etoposide IV continuously over 96 hours beginning on day 1 and continuing until day 5, and filgrastim (G-CSF) subcutaneously (SC) daily beginning on day 6 and continuing until day 19 or until blood counts recover OR pegfilgrastim SC on day 6.

NOTE: *Patients may receive iCDE without bevacizumab if they meet any exclusion criteria for receiving bevacizumab.

Treatment with bevacizumab and iCDE repeats every 21 days for 4-8 courses in the absence of disease progression or unacceptable toxicity. Patients achieving complete response (CR) receive 2 additional courses beyond CR.

After completion of study treatment, patients are followed monthly for 6 months, every 2 months for 6 months, every 3 months for 1 year, every 6 months for 3 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 15 patients will be accrued for this study within 2.5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed primary effusion lymphoma (PEL) involving a body cavity

  * Kaposi's sarcoma associated-herpesvirus
  * Any anatomic site or distribution of involvement allowed
  * HIV infection allowed
* Previously treated or untreated disease
* No mass lesions in the brain (for patients receiving bevacizumab during study treatment)

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-3* NOTE: *ECOG 4 allowed if due to a mechanical effect of the PEL that can be corrected by effusion drainage resulting in improved performance status to ECOG 3 or better

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count > 1,000/mm^3
* Platelet count > 75,000/mm^3
* No active bleeding or coagulopathy (for patients receiving bevacizumab during study treatment)

Hepatic

* AST and ALT < 3 times upper limit of normal (ULN) (6 times ULN if due to hyperalimentation)
* Bilirubin < 2.0 mg/dL OR
* Total bilirubin ≤ 4.5 mg/dL AND direct bilirubin < 0.4 mg/dL (for patients with Gilbert's syndrome or receiving protease-inhibitor therapy)

Renal

* Creatinine ≤ 1.5 mg/dL OR
* Creatinine clearance > 50 mL/min

Cardiovascular

* Patients receiving bevacizumab during study treatment must meet the following criteria:

  * No deep venous or arterial thrombosis within the past 6 months
  * No uncontrolled hypertension (i.e., systolic blood pressure [BP] > 160 mm Hg or diastolic BP > 95 mm Hg)
  * No unstable angina
  * No New York Heart Association class II-IV congestive heart failure
  * No cardiac arrhythmia requiring medication
  * No clinically significant peripheral artery disease
  * No peripheral vascular disease ≥ grade 2
  * No prior myocardial infarction
  * No transient ischemic attack or cerebral vascular accident within the past 6 months
  * No other clinically significant cardiovascular disease

Neurologic

* Patients receiving bevacizumab during study treatment must meet the following criteria:

  * No uncontrolled seizure disorder
  * No CNS bleeding within the past 6 months
  * No other substantial CNS disease

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No other malignancy requiring treatment that would preclude study treatment, including, but not limited to, any of the following:

  * Life-threatening Kaposi's sarcoma
  * Non-resectable lung cancer
  * Acute leukemia
* No grade IV organ dysfunction unrelated to PEL
* No infection requiring chronic systemic therapy that would preclude study treatment (except HIV, hepatitis B, or hepatitis C), including, but not limited to, any of the following:

  * Invasive aspergillosis
  * End-organ cytomegalovirus (CMV)

    * CMV retinitis (e.g., ocular implants not requiring systemic therapy) allowed if controlled with local therapy
* No other condition or circumstance that would preclude study participation
* No gastrointestinal bleeding within the past 6 months (for patients receiving bevacizumab during study treatment)
* No pathological condition that would confer a high risk for bleeding (for patients receiving bevacizumab during study treatment)

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No live virus vaccines (e.g., vaccinia or rotavirus) or bacterial vaccines during and for 3 months after completion of study treatment

Chemotherapy

* No prior cumulative anthracycline dose > 450 mg/m^2 (unless cardiac ejection fraction normal)

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Other

* No concurrent chronic daily aspirin ≥ 325 mg/day or nonsteroidal medication that interferes with platelet function (for patients receiving bevacizumab during study treatment)
* No concurrent therapeutic anticoagulation (INR > 1.5) unless patient is on full-dose warfarin (for patients receiving bevacizumab during study treatment)

  * Full-dose anticoagulants allowed provided both of the following criteria are met:

    * INR normal
    * On a stable dose of warfarin or low-molecular weight heparin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2005-07; Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Response to therapy as measured by overall, disease-free, and progression-free survival each month

SECONDARY OUTCOMES:
Effects of high-dose zidovudine and ganciclovir on tumor cells measured by various assays after 2 weeks of study treatment

CONTACTS AND LOCATIONS:
Overall Officials: Richard F. Little, MD, Principal Investigator — NCI - HIV and AIDS Malignancy Branch
Locations (1):
- Warren Grant Magnuson Clinical Center - NCI Clinical Trials Referral Office, Bethesda, Maryland, United States